CLINICAL TRIAL: NCT04793152
Title: Vancomycin Dosing for Serious MRSA Infections: A Non-inferiority Randomized Trial of Trough Level Versus AUC/MIC
Acronym: TAUC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anthony Bai (Other)
Collaborators: Physician Services Incorporated (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Anthony Bai, Assistant Professor - Dept of Medicine, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13327
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: MRSA
Keywords: vancomycin; MRSA; trough; AUC
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vancomycin targeting trough of 10 to 15mg/L (Experimental): If the patient has not received intravenous vancomycin yet, a loading dose of 25mg/kg (maximum 2g) will be given if the patient is severely ill at the discretion of the physician and pharmacist. The initial dose is 15mg/kg with a maximum dose of 2g. The frequency would be based on creatinine clearance (CrCl) as per the Cockcroft-Gault equation: Q8H if CrCl is >100mL/min, Q12H if CrCl is 50-100mL/min, Q24H if CrCl is 30- 49mL/min, and Q48H if CrCl is <30mL/min. Pharmacists can change the initial dose at their own discretion.
  Trough level will be done 30 minutes before the 4th dose. For Q48H dosing, a trough level will be done before the second dose. Vancomycin dosing will be adjusted to target trough level of 10 to 15mg/L. If not at target, the pharmacist will adjust the dose based on an assumption of linear pharmacokinetics. Trough will be remeasured before the fourth dose of the new regimen.
  Interventions: Drug: Vancomycin
- Vancomycin targeting AUC of 400 to 600 (Active Comparator): The initial intravenous vancomycin dosing is the same as described above for the trough group.
  The AUC target will be 400 to 600, which assumes a MIC of 1ug/mL by broth microdilution.
  After the first non-loading dose of vancomycin, patients will have vancomycin level 30 minutes before the next dose. As per the pharmacist's discretion, patient may have an additional vancomycin level one hour after infusion of vancomycin for more accurate estimates. A pharmacist will use a Bayesian software to estimate the AUC and the optimal dose.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Administration as outlined

SUMMARY:
Intravenous vancomycin is considered first line therapy for serious methicillin-resistant Staphylococcus aureus (MRSA) infections including bacteremia, central nervous system infection, pneumonia, pleural space infection, bone or joint infection, prosthetic joint infection and deep abscesses. The effectiveness and toxicity of vancomycin depend on its dosing and chosen target. The most recent guidelines suggest targeting area under the curve over 24 hours over minimum inhibitory concentration (AUC/MIC) of 400 to 600. Implementation of AUC/MIC requires Bayesian software that can be variable, costly, complicated and time consuming. Ideally, AUC/MIC dosing would also require susceptibility testing by broth microdilution, which is not commonly done. It is recommended to target AUC of 400 to 600 assuming a MIC of 1ug/mL when MIC by broth microdilution is not known. Targeting a trough level of 10 to 15mg/L may be a reasonable and more practical alternative without compromising effectiveness. We will be conducting a randomized controlled non-inferiority trial to compare intravenous vancomycin dosing strategy targeting a trough level of 10 to 15mg/L versus AUC of 400 to 600 assuming a MIC of 1ug/mL by broth microdilution for serious MRSA infections. The primary outcome will be treatment failure, which is a composite of mortality and microbiologic failure at 90 days. We hypothesize that targeting a trough level of 10 to 15mg/L is non-inferior to targeting a AUC of 400 to 600 in terms of treatment failure. The criterion for non-inferiority is that a two-sided 95% confidence interval for difference in risk of treatment failure will lie within the non-inferiority margin of 10%.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with serious MRSA infections based on culture results including bacteremia, pneumonia, pleural space infection, central nervous system infection, bone infection, septic arthritis, prosthetic joint infection, and deep abscess
* Enrolment within 4 days from date of MRSA culture collection
* Patient either currently not on vancomycin or has received vancomycin for 4 days or less

Exclusion Criteria:

* Vancomycin minimum inhibitory concentration (MIC) ≥2ug/mL
* Patient is palliative or expected to die in the next 48 hours, or requires critical care resources but will not receive it due to advanced care directives
* History of type 1 hypersensitivity reaction to vancomycin
* Patients on intermittent hemodialysis or peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 90 days
  Treatment failure is defined as death due to any cause or microbiologic failure based on demonstration of MRSA on repeated culture from the original site or another sterile site more than 1 week from randomization. Treatment failure will be determined by an independent committee of physicians after reviewing the clinical, laboratory and microbiologic data.

SECONDARY OUTCOMES:
Major adverse kidney events | 90 days
  New and persistent renal-replacement therapy, or serum creatinine that is 200% or more than the baseline value during the follow-up period
Vancomycin associated nephrotoxicity | 90 days
  Increase in serum creatinine by ≥26.4mmol/L or ≥50% since starting vancomycin when compared to baseline
Renal replacement therapy | 90 days
  Need for initiation of renal replacement therapy at any time during follow-up
Time to target | 90 days
  Time in days to reach target level (trough of 10 to 15mg/L in the intervention group and AUC/MIC of 400 to 600 in the comparison group)
Day 3 AUC | 3 days
  AUC as calculated using Bayesian modeling on day 3 from randomization
Vancomycin cost | 90 days
  Direct cost of vancomycin monitoring and dosing from perspective of hospital system

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Bai, MD, Principal Investigator — Queen's University
Locations (4):
- Canada (4):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No